CLINICAL TRIAL: NCT04053582
Title: Augmented Mindfulness Training for Resilience in Early Life
Acronym: A-MindREaL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LIBR # 2019-003-01; 5P20GM121312 (NIH)
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Adolescents With Early Life Stress
Keywords: Early life adversity; Adolescents; Mindfulness; Neurobiology; Stress and resilience
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: ELA-exposed youth are randomly assigned to receive augmented mindfulness training with real-time neurofeedback or a sham condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented Mindfulness Training (AMT) (Active Comparator): Participants will receive real-time neurofeedback from the PCC during mindfulness practice in the MRI
  Interventions: Behavioral: AMT
- Sham (Active Comparator): Participants will receive an artificial neurofeedback signal during mindfulness practice in the MRI
  Interventions: Behavioral: Sham

INTERVENTIONS:
Behavioral: AMT — The session will be done on an individual basis. AMT group will receive neurofeedback training from the PCC while focusing on the physical sensations of the breath. The session will last one hour, including 3 neurofeedback runs during which subjects will undergo three conditions across three consecutive blocks: Rest (30s), Describe (view an adjective and decide whether the word describes them; 20s), and Focus on the Breath with neurofeedback (70s).
  Arms: Augmented Mindfulness Training (AMT)
Behavioral: Sham — The session will be done on an individual basis. Sham group will receive artificial neurofeedback while focusing on the physical sensations of the breath. The session will last one hour, including 3 sham neurofeedback runs during which subjects will undergo three conditions across three consecutive blocks: Rest (30s), Describe (view an adjective and decide whether the word describes them; 20s), and Focus on the Breath with artificial neurofeedback (70s).
  Arms: Sham

SUMMARY:
This project aims to determine whether neurofeedback augmented mindfulness intervention increases the plasticity in brain areas affected by exposure to early life adversity in youth. The study will first establish the augmented mindfulness training protocol targeting the posterior cingulate cortex (PCC) with real-time fMRI neurofeedback for use with healthy control and ELA-exposed youth. Next, in addition to ongoing data collection with healthy controls, ELA-exposed youth will be randomly assigned to either complete the neurofeedback augmented mindfulness training (AMT) or sham condition protocol. Effect of augmented mindfulness training on state measures of mindfulness, perceived stress, and affect will be examined.

DETAILED DESCRIPTION:
Early life adversity (ELA) is a major public health crisis that results in significant disruptions in neurobiological processes and long-term psychiatric and health consequences, yet very little is known about interventions that may prevent them and the optimal time to do so. Not only is ELA associated with earlier onset and greater severity and comorbidity of depression, anxiety, and substance abuse, these individuals also evidence significantly poorer responses to psychological and pharmacological interventions when treated for these conditions. Consequently, there is a dire need to develop preventive interventions that target individuals with ELA exposure. The first step in this process is to establish malleability of neural mechanisms disrupted by ELA exposure to acute interventions. We use augmented mindfulness training, that is, a standard mindfulness training combined with real-time functional magnetic resonance imaging neurofeedback (rtfMRI-nf) to influence and increase the plasticity of brain areas affected by ELA, in turn affecting state changes in symptoms in youth with ELA exposure. These fMRI tasks are designed to engage the PCC and mindfulness practice.

Over the course of three years, 120 eligible youth with early life adversity or healthy controls will be recruited into the study. All healthy controls will receive AMT, and ELA-exposed youth will be randomly assigned to AMT, consisting of real-time fMRI with neurofeedback during mindfulness practice, or Sham, consisting of artificially calculated neurofeedback signals during mindfulness practice. Adolescents will complete self-report measures to assess state affective symptoms before and after receiving mindfulness training and scanning, and again one week later.

ELIGIBILITY:
Inclusion criteria:

Healthy controls (n=48):

* Age 13.00 - 17.99 years at time of baseline assessment
* Able to validly and safely complete baseline assessments
* All genders
* All races

ELA-exposed participants (n=72):

* Age 13.00 - 17.99 years at time of baseline assessment
* Able to validly and safely complete baseline assessments
* All genders
* All races
* Endorsing 4 or more types of maltreatments on the Maltreatment and Abuse Chronology and Exposure (MACE) scale, OR meeting the cutoff score on 2 or more of the 5 subscales on the Childhood Trauma Questionnaire (CTQ):

Sexual abuse ≥ 8 Physical abuse ≥ 8 Emotional abuse ≥ 10 Physical neglect ≥ 8 Emotional neglect ≥ 15

* Moderate levels of depression or anxiety (one standard deviation above the mean) as measured by the NIH PROMIS measures

Exclusion criteria:

All participants:

* No biological parent or legal guardian identified to give permission for minor to participate
* History of neurological disorders including seizure disorder, cerebral palsy, or other conditions requiring neurological or medical care, being managed for migraines (e.g., daily prophylactic medication, seeing a neurologist for migraines), or a diagnosis of Developmental Delay, including severe learning disorder, mental retardation, autism spectrum disorders, pervasive developmental disorder, or other conditions requiring repeated and persistent specialized education.
* Current psychotic disorder, bipolar disorder, obsessive-compulsive and related disorders, substance use disorder, conduct problems (i.e., conduct or oppositional defiant disorder).
* Current use of medications with major effects on brain function or blood flow (e.g., antipsychotics, acne medications). For ELA-exposed participants, the use of one (1) medication (e.g., SSRI's, ADHD medications) will not be exclusionary permitting that participant has been on a stable dosage for at least 6 weeks prior to study enrollment.
* MRI contraindications including: cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a professional metal worker/welder, history of eye surgery/eyes washed out because of metal, vision problems uncorrectable with lenses, inability to lie still on one's back for 60-120 minutes; prior neurosurgery; tattoos or cosmetic makeup with metal dyes, unwillingness to remove body piercings, and pregnancy
* Unwillingness or inability to complete any of the major aspects of the study protocol, including magnetic resonance imaging (i.e., due to claustrophobia) or behavioral assessment. However, failing to complete some individual aspects of these assessment sessions will be acceptable (i.e., being unwilling to answer individual items on some questionnaires).
* Severe claustrophobia
* Not fluent in English
* Weight less than 100 lbs.
* Non-correctable vision, hearing or sensorimotor impairments, as protocol elements may not be valid
* Youth planning to move to an area not within reasonable traveling distance of LIBR; knowledge at baseline that treatment completion/follow-up will not be possible
* Youth appears to be high/intoxicated, or withdrawing from the effects of alcohol or drugs at time of enrollment

Healthy controls:

* History of or current psychiatric illness
* Endorsing 2 or more types of maltreatments on the Maltreatment and Abuse Chronology and Exposure (MACE) scale, or meeting the cutoff score on one or more of the subscales on the Childhood Trauma Questionnaire (CTQ) Sexual abuse ≥ 8 Physical abuse ≥ 8 Emotional abuse ≥ 10 Physical neglect ≥ 8 Emotional neglect ≥ 15
* Current use of medications with major effects on brain function or blood flow (e.g., antipsychotics, mood stabilizers, ADHD medications, SSRIs, and acne medications).

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Percent signal change in the Posterior Cingulate Cortex (PCC) as assessed by fMRI | Through study completion (average: 2 weeks)
  Percent signal change in the PCC for Focus - Describe condition contrast will be lower in the AMT relative to the Sham group during mindfulness practice.

SECONDARY OUTCOMES:
State Mindfulness Scale (SMS) scores | Through study completion (average: 2 weeks)
  The SMS is a 21-item measure rated on a 5-point Likert scale (not at all - very well). Items may be summed or averaged, with greater scores indicating greater levels of state mindfulness. SMS scores will evidence a greater increase from pre- to post-training and 1-week follow-up in the AMT relative to the Sham group.
Perceived Stress Scale (PSS) scores | Through study completion (average: 2 weeks)
  The PSS is a 10 item measure on a 5-point Likert scale (never - very often), with 4 items reverse scaled. Items are summed, with greater scores indicating greater levels of perceived stress. PSS scores will evidence a greater decrease from pre- to post-training and 1-week follow-up in AMT relative to the Sham group.
Positive and Negative Affect Schedule for Children (PANAS-C) scores | Through study completion (average: 2 weeks)
  The PANAS-C assesses domains of positive and negative affect on a 5-point Likert scale (not much or not at all - a lot) with 30 items. Scores for each domain are summed, with greater scores indicating greater levels of its respective affective domain. PANAS-C scores will evidence a greater change from pre- to post-training and 1-week follow-up in AMT relative to the Sham group.

CONTACTS AND LOCATIONS:
Overall Officials: Namik Kirlic, PhD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cosgrove KT, Tsuchiyagaito A, Cohen ZP, Cochran G, Yu X, Misaki M, Aupperle RL, Singh MK, Paulus MP, Kirlic N. Augmenting mindfulness training through neurofeedback: a pilot study of the pre-post changes on resting-state functional connectivity in typically developing adolescents. Front Neurosci. 2024 Oct 30;18:1397234. doi: 10.3389/fnins.2024.1397234. eCollection 2024. PMID 39539491
- [Derived] Kirlic N, Cohen ZP, Tsuchiyagaito A, Misaki M, McDermott TJ, Aupperle RL, Stewart JL, Singh MK, Paulus MP, Bodurka J. Self-regulation of the posterior cingulate cortex with real-time fMRI neurofeedback augmented mindfulness training in healthy adolescents: A nonrandomized feasibility study. Cogn Affect Behav Neurosci. 2022 Aug;22(4):849-867. doi: 10.3758/s13415-022-00991-4. Epub 2022 Mar 15. PMID 35292905

DOCUMENTS (1):
  • Informed Consent Form (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT04053582/ICF_000.pdf